CLINICAL TRIAL: NCT06881992
Title: A Phase 3, Single-Arm, Open-label, Pivotal Study to Evaluate the Efficacy and Safety of Ersodetug Compared to Baseline in Patients With Inadequately Controlled Hypoglycemia Due to Tumor Hyperinsulinism (Tumor HI)
Brief Title: A Phase 3 Study of Ersodetug in Patients With Tumor Hyperinsulinism
Acronym: Tumor HI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rezolute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RZ358-302
Record Dates: First submitted 2025-03-10; First posted 2025-03-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Tumor Hyperinsulinism (Tumor HI)
Keywords: Doege-Potter Syndrome; Ectopic insulinoma; Extra-pancreatic insulinoma; Fibrosarcoma; HCC; Hyperinsulinemia; Hypoglycemia; Hypoglycemia due to fibrosarcoma; Hypoglycemia due to HCC; Hypoglycemia due to liposarcoma; Hypoglycemia due to tumor/cancer; IGF 2 Insulinoma; IGF 2 mediated non islet cell tumor hypoglycemia; IGF-2 mediated hypoglycemia; IGF-2, Big IGF-2; IGF-oma, IGF-2-oma, Big IGF-2-oma; Insulinoma; Islet cell tumor (ICT); Liposarcoma; Neuroendocrine tumor (NET); NICTH; Non Islet Cell Tumor; Non-islet cell tumor hypoglycemia (NICTH); Paraneoplastic; Paraneoplastic hypoglycemia; PNET; Pro-insulinoma; Tumor/cancer associated hypoglycemia; Tumor/cancer induced hypoglycemia; Tumor/cancer mediated hypoglycemia; Clinical Trials for: -Insulinoma -proinsulinoma -extrapancreatic insulinoma -non-islet cell tumor -IGF-oma -HCC -Liposarcoma -Fibrosarcoma
MeSH Terms: conditions — Fibrosarcoma; Hyperinsulinism; Hypoglycemia; Neoplasms; Insulinoma; Adenoma, Islet Cell; Liposarcoma; Neuroendocrine Tumors; Neuroectodermal Tumors, Primitive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with a diagnosis of Tumor HI (insulin- or IGF-producing tumors) (Other)
  Interventions: Drug: Ersodetug

INTERVENTIONS:
Drug: Ersodetug — Ersodetug (9 mg/kg) + SOC

SUMMARY:
The objectives of this study are to evaluate the glycemic efficacy, safety, and tolerability of ersodetug as add-on to standard of care (SOC) therapy for treatment of hypoglycemia in patients with Tumor Hyperinsulinism (Tumor HI).

DETAILED DESCRIPTION:
This study will include participants who are suffering from low blood sugar related symptoms (hypoglycemia) due to over-production of hormones (e.g. insulin or similar substances) by certain non-removable tumors that cannot be treated satisfactorily with available treatment. Every study participant will receive ersodetug doses weekly for 8 weeks alongside their usual treatments for hypoglycemia at a dose of 9 mg/kg.

The study is divided into 3 periods: Screening (up to 4 weeks), Treatment (8 weeks) and either End of Study Follow-up (approximately up to 20 weeks after the last dose) or optional Open Label Extension (OLE) phase (up to 3 years).

This study is being conducted at approximately 10-15 study sites in approximately 5 countries. The study will enroll approximately 16 participants, all with a diagnosis of tumor HI (insulin- or IGF producing tumors).

ELIGIBILITY:
Inclusion Criteria:

* The eligibility criteria of all participants must be evaluated by a multidisciplinary team led by the PI, which must include an oncologist
* Male or female participants of ≥18 years of age who provide written informed consent.
* Clinical diagnosis of neuroendocrine tumor (NET) (ICT or NICT) with biochemical evidence of tumor hyperinsulinism (hypoglycemia with inappropriately elevated insulin or insulin-like growth factor (IGF)/variant suppression) confirmed via laboratory assessment who have failed to achieve adequate control of hypoglycemia with usual SOC anti-hypoglycemic therapies, per investigator judgement.
* Currently requiring IV glucose infusion and/or parenteral nutrition for ≥7 days for the management of refractory hypoglycemia (prior to administration of the 1st dose of ersodetug).

Exclusion Criteria:

* Evidence of active infection including human immunodeficiency virus, hepatitis B, or hepatitis C (excluding immunization patterns).
* Treatment with an investigational drug or device within 30 days or 5 half-lives of the investigational drug (whichever is longer), however, if the treating physician and Medical Monitor consider no significant risk of drug-drug interaction and potential benefit outweighs the risk then the participant may be allowed to participate. Participation in registries and purely diagnostic studies is allowed
* Any out-of-range laboratory value at screening (other than glucose) that is assessed as clinically significant by the investigator. Laboratory or radiographic abnormalities that are considered related to the underlying disease (tumor) or associated therapies and do not pose additional safety risk for study participation per investigator and Medical Monitor may be allowed.
* Known allergy or sensitivity to ersodetug or any component of the drug.
* Any organ condition, concomitant disease (e.g., psychiatric illness, severe alcoholism, or drug abuse, cardiac, hepatic, or kidney disease), or other abnormality that itself, or the treatment of which in the opinion of the investigator and/or Sponsor's Medical Monitor would pose an unacceptable risk to the participant in the study.
* Estimated life expectancy (additional lifespan) due to underlying disease (tumor) is <8 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with clinically meaningful reduction in IV glucose infusion rate from baseline. | 8 weeks

SECONDARY OUTCOMES:
Change from baseline in average daily IV glucose/dextrose infusion rate (GIR). | 8 weeks
Change from baseline in average daily total IV glucose delivery (g) | 8 weeks
Time to complete weaning off IV glucose administration after initiating ersodetug. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (13):
- United States (8):
  - Investigative Site, Chicago, Illinois
  - Investigative Site, Bethesda, Maryland
  - Investigative Site, Boston, Massachusetts
  - Investigative Site, Rochester, Minnesota
  - Investigative Site, New York, New York
  - Investigative Site, Canton, Ohio
  - Investigative Site, Portland, Oregon
  - Investigative Site, Houston, Texas
- Investigative Site, Clichy, Île-de-France Region, France
- Investigative Site, Rotterdam, South Holland, Netherlands
- Investigative Site, Basel, Canton Basel-Stadt, Switzerland
- United Kingdom (2):
  - Investigative Site, Saint Johns Wood, London
  - Investigative Site, Withington, Manchester